CLINICAL TRIAL: NCT05394116
Title: Phase 3 Randomized, Placebo-Controlled Study to Assess Safety, Tolerability, and Efficacy of Garetosmab in Patients With Fibrodysplasia Ossificans Progressiva
Brief Title: A Study to Assess Safety, Tolerability and Efficacy of Garetosmab Versus Placebo Administered Intravenously (IV) in Adult Participants With Fibrodysplasia Ossificans Progressiva (FOP)
Acronym: OPTIMA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R2477-FOP-2175; 2022-000880-40 (Registry Identifier: EudraCT); 2023-508350-26-00 (Registry Identifier: CTIS (EU))
Expanded Access: NCT07301450 (Temporarily not available)
Record Dates: First submitted 2022-05-04; First posted 2022-05-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Fibrodysplasia Ossificans Progressiva
Keywords: Heterotopic Ossification (HO) Lesions; Type I activin A receptor (ACVR1); Optima; LUMINA-1; Flare-Ups
MeSH Terms: conditions — Myositis Ossificans; Ossification, Heterotopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High dose Garetosmab (Experimental): Garetosmab is administered by intravenous (IV) administration every 4 weeks (Q4W)
  Interventions: Drug: Garetosmab
- Low dose Garetosmab (Experimental): Garetosmab is administered by IV administration Q4W
  Interventions: Drug: Garetosmab
- Placebo (Experimental): Placebo to match garetosmab, is supplied as a liquid solution without the monoclonal antibody (or the protein) and is administered IV Q4W.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Garetosmab — Garetosmab is supplied as a liquid drug product and will be administered IV.
  Other Names: REGN2477
  Arms: High dose Garetosmab; Low dose Garetosmab
Drug: Placebo — Placebo to match garetosmab, is supplied as a liquid solution without the monoclonal antibody (or the protein) and is administered IV.
  Arms: Placebo

SUMMARY:
This study is researching an experimental drug called garetosmab. The study is focused on adult patients with fibrodysplasia ossificans progressiva (FOP).

The aim of the study is to see how safe and effective the study drug is in patients with FOP.

The study is looking at several other research questions, including:

* What side effects may happen from receiving the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Clinical diagnosis of Fibrodysplasia Ossificans Progressiva (FOP) [(based on findings of congenital malformation of the great toes, episodic soft tissue swelling, and/or progressive Heterotopic Ossification (HO)]
2. Confirmation of FOP diagnosis with documentation of Type I activin A receptor (ACVR1) FOP causing mutation
3. FOP disease activity within 1 year of screening visit. FOP disease activity is defined as pain, swelling, stiffness, or other signs and symptoms associated with FOP flare-ups; or worsening of joint function, or radiographic progression of HO lesions (increase in size or number of HO lesions) with/without being associated with flare-up episodes
4. Willing and able to undergo CT imaging procedures and other procedures as defined in the protocol

Key Exclusion Criteria:

1. Cumulative Analog Joint Involvement Scale (CAJIS) score at screening >19
2. Participant has significant concomitant illness or history of significant illness such as but not limited to cardiac, renal, rheumatologic, neurologic, psychiatric, endocrine, metabolic, or lymphatic disease, that in the opinion of the study investigator might confound the results of the study or pose additional risk to the patient by their participation in the study
3. Previous history or diagnosis of cancer
4. Severely impaired renal function defined as estimated glomerular filtration rate <30 milliliter per minute (mL/min) (/1.73 m^2 calculated by the Modification of Diet in Renal Disease equation
5. Uncontrolled diabetes defined as hemoglobin A1C (HbA1c) >9% at screening
6. History of poorly controlled hypertension, as defined by:

   1. Systolic blood pressure ≥180 mm Hg or diastolic blood pressure ≥110 mm Hg at the screening visit
   2. Systolic blood pressure of 160 mm Hg to 179 mm Hg or diastolic blood pressure of 100 mm Hg to 10^9 mm Hg at the screening visit, AND a history of end-organ damage (including history of left-ventricular hypertrophy, heart failure, angina, myocardial infarction, stroke, transient ischemic attack, peripheral arterial disease, end-stage renal disease, and moderate-to-advanced retinopathy
7. Known history of cerebral vascular malformation
8. Cardiovascular conditions such as New York Heart Association class III or IV heart failure, cardiomyopathy, intermittent claudication, myocardial infarction, or acute coronary syndrome within 6 months prior to screening; symptomatic ventricular cardiac arrhythmia
9. History of severe respiratory compromise requiring oxygen, respiratory support (eg, bilevel positive airway pressure [biPAP] or continuous positive airway pressure [CPAP]), or a history of aspiration pneumonia requiring hospitalization
10. Prior use in the past year and concomitant use of bisphosphonates
11. Concurrent participation in another interventional clinical study or a non-interventional study with radiographic measures or invasive procedures (eg, collection of blood or tissue samples)
12. Treatment with another investigational drug, denosumab, imatinib or isotretinoin in the last 30 days or within 5 half-lives of the investigational drug, whichever is longer
13. Pregnant or breastfeeding women
14. Women of childbearing potential (WOCBP) who are unwilling to practice highly effective contraception, as defined in the protocol
15. Male patients with WOCBP partners who are not willing to use condoms with WOCBP partners to prevent potential fetal exposure, as defined in the protocol

Note: Other protocol defined Inclusion/Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2029-02-27 (Estimated)

PRIMARY OUTCOMES:
Number of new HO lesions | At Week 56
Incidence and severity of treatment-emergent adverse events of special interest (AESIs) | Baseline to Week 56

SECONDARY OUTCOMES:
Number of clinician-assessed flare-ups | Through Weeks 28, 56 and 84
  Investigator assess flare-up events according to his/her medical judgment. A FOP flare-up is characterized as episodic, painful inflammatory soft tissue swelling.
  Week 84 Only for Patients on Extended Treatment
Occurrence of new HO lesions | At Weeks 28, 56 and 84
  Reported as Yes/No
  Week 84 Only for Patients on Extended Treatment
Total volume of new HO lesions | At Weeks 28, 56 and 84
  Week 84 Only for Patients on Extended Treatment
Occurrence of patient-reported flare-ups | Through Weeks 28 and 56
  Reported as Yes/No
Number of new HO lesions | At week 28 and 84
  Week 84 Only for Patients on Extended Treatment
Occurrence of clinician-assessed flare-ups | Through Weeks 28, 56 and 84
  Reported as Yes/No
  Week 84 Only for Patients on Extended Treatment
Number of patient-reported flare-ups | Through Weeks 28 and 56
  Flare-up is defined as two or more of the following: pain, swelling, joint stiffness, or decrease in movement. The FOP flare-up dairy is a questionnaire and is self-completed by the participant daily.
Change in joint function assessment by physician using cumulative analog joint involvement scale (CAJIS) | Baseline to Weeks 28 and 56
  CAJIS is a clinician assessment of 15 major joints; each major joint rated normal unaffected (0), affected (1), or completely functionally ankylosed (2). The total score ranges from 0 to 30
Change in pulmonary function as assessed by spirometry | Baseline at Weeks 28 and 56
  Forced vital capacity (FVC) and Forced expiratory volume in 1 second (FEV1) and the ratio of FEV1/FVC will be determined by spirometry.
Change in disease severity as assessed by the Patient Global Impression of Severity (PGIS) | Baseline to Weeks 28 and 56
  PGIS is a single item, self-administered questionnaire to assess the patient's global impression of severity
Change in disease severity as assessed by the Patient's Global Impression of Change (PGIC) | At Weeks 28 and 56
  PGIC is a single item, self-administered questionnaire to assess the patient's global impression of change
Change in disease severity as assessed by the Clinician's Global Impression of Change (CGIC) | At Weeks 28 and 56
  CGIC is a single-item questionnaire to assess the clinician's global impression of change
Concentration of total activin A in serum over time | Through Week 56
Concentration of garetosmab in serum over time | Through Week 56
Incidence of anti-drug antibodies (ADA) to garetosmab over time | Through Week 56
Titer of ADA to garetosmab over time | Through Week 56

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (22):
- United States (2):
  - University of California Los Angeles (UCLA) Medical Center, Los Angeles, California
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Royal North Shore Hospital, St Leonards, New South Wales, Australia
- Hospital Israelita Albert Einstein, São Paulo, Brazil
- Universidad de Concepcion, Concepción, Bio Bio, Chile
- Tongji Hospital of Tongji University, Shanghai, China
- Clinica Universidad de La Sabana, Chía, Cundinamarca, Colombia
- HUS Children and Adolescents Park Hospital Clinical Trial Unit, Helsinki, Stenbäckinkatu 11, Finland
- France (2):
  - Hôpital Lapeyronie, Montpellier
  - Hopital Lariboisiere, Paris
- Queen Mary Hospital, Hong Kong, Hong Kong
- IRCCS Istituto Giannina Gaslini, Genoa, Italy
- Japan (3):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Oita University Hospital, Yufu, Oita Prefecture
  - Kyushu University Hospital, Fukuoka
- Hospital Kuala Lampur, Kuala Lumpur, Malaysia
- Amsterdam University Medical Center, Amsterdam, North Holland, Netherlands
- Szpital Centrum Medyczne Medyk, Rzeszów, Podkarpackie Voivodeship, Poland
- University of Cape Town, Rondebosch, Cape Town, South Africa
- Seoul National University Hospital, Seoul, South Korea
- Hospital Universitario Ramon y Cajal, Madrid, Spain
- Royal National Orthropaedic Hospital NHS Trust, Middlesex, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/